CLINICAL TRIAL: NCT02550886
Title: Anticipated Versus Actual Patient and Caregiver Burden Following Ambulatory Orthopedic Surgery
Acronym: Work Burden
Status: Terminated | Type: Observational
Why Stopped: Lost many participants to follow-up.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-395
Record Dates: First submitted 2015-08-31; First posted 2015-09-16 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Stress, Psychological; Pain
Keywords: Work Burden; Ambulatory Orthopedic Surgery; Anesthesiology; Perioperative Care
MeSH Terms: conditions — Stress, Psychological; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient/Caregiver Dyad
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients and their caregivers will be asked to complete surveys about their expected and actual time taken off from work. They will also answer questions about the patient's recovery, as well as the patient/caregiver relationship.

SUMMARY:
In 2011, 38.6 million hospital stays occurred in the United States at a cost of $387.2 billion. 47.9 percent involved hospitalizations during which surgical procedures were performed. Orthopedic procedures constituted the most frequently performed and most costly of operating room procedures. As the healthcare climate in the United States continues to change, there is a trend towards providing effective care in a fiscally conservative manner. Central to this strategy is the shift towards increasing ambulatory surgical procedures from surgeries requiring post-operative admission for patients. While savings to hospitals and third-party payers are implied, there may be an unrecognized increase in financial, physical, and psychosocial post-operative costs to patients undergoing ambulatory surgery and to their caregivers. Rawal et al., and McGarth and colleagues have found that patients undergoing orthopedic procedures had moderate to severe post-operative pain. We propose to present a survey to patients and their caregivers before surgery and at multiple timepoints post-operatively to acquire information on the impacts of ambulatory orthopedic surgery. In addition to assessing post-operative pain, this study serves to examine various other possible burdens to patients that have not been previously evaluated in this patient population.

REFERENCES

McGarth B, Elgendy H, Chung F, Kamming D, Curti B, King S. Thirty percent of patients have a moderate to severe pain 24 hr after ambulatory surgery: a survey of 5,703 patients. Can J Anesth. 2004; 51:886-891.

Rawal N, Hylander J, Nydahl P, Olofsson I, Gupta A. Survey of postoperative analgesia following ambulatory surgery. Acta Anesthesiol Scand. 1997; 41:1017-1022.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing outpatient arthroscopic knee debridement or meniscectomy surgery
* Age 18-85
* Primary caregiver available during preoperative period who is employed full-time or part-time
* English speaking
* Patients who are employed full-time or part-time

Exclusion Criteria:

* Patients on disability or worker's compensation
* Patients undergoing concurrent procedures
* Patients who are self-employed
* Caregivers who are self-employed
* Surgeons: Dr. Altchek, Dr. Warren, Dr. O'Brien

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing outpatient arthroscopic knee debridement or meniscectomy surgery at Hospital for Special Surgery
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Time taken off from work--specifically, the number of extra days taken off from work by patients and their caregivers after surgery | Holding area before surgery, post-operative day 1 (POD 1), POD 7, biweekly thereafter until patient returns to baseline level of work, and two weeks after patient returns to baseline level of work
  Patients and caregivers will be considered able to return to their baseline level of work once they can fulfill all responsibilities at their current occupation with no restrictions.

SECONDARY OUTCOMES:
Expected Burden of Recovery | Holding area before surgery, post-operative day 1 (POD 1), POD 7, biweekly thereafter until patient returns to baseline level of work, and two weeks after patient returns to baseline level of work
  1. Patient: pain, nausea, vomiting, doctor appointments/hospital visits, days to return to daily activities, days to achieve recovery, days missed from work, emotional duress
  2. Caregiver: days missed from work; days to return to daily activities; emotional duress; productivity, sleep, work and personal adjustments
Excess (Actual Beyond Expected) Burden of Recovery | Holding area before surgery, post-operative day 1 (POD 1), POD 7, biweekly thereafter until patient returns to baseline level of work, and two weeks after patient returns to baseline level of work
  1. Patient: pain, nausea, vomiting, doctor appointments/hospital visits, days to return to daily activities, days to achieve recovery beyond expected, days missed from work, emotional duress
  2. Caregiver: days missed from work; days to return to daily activities; emotional duress; productivity, sleep, work and personal adjustments

CONTACTS AND LOCATIONS:
Overall Officials: Kanupriya Kumar, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery (HSS), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGrath B, Elgendy H, Chung F, Kamming D, Curti B, King S. Thirty percent of patients have moderate to severe pain 24 hr after ambulatory surgery: a survey of 5,703 patients. Can J Anaesth. 2004 Nov;51(9):886-91. doi: 10.1007/BF03018885. PMID 15525613
- [Background] Rawal N, Hylander J, Nydahl PA, Olofsson I, Gupta A. Survey of postoperative analgesia following ambulatory surgery. Acta Anaesthesiol Scand. 1997 Sep;41(8):1017-22. doi: 10.1111/j.1399-6576.1997.tb04829.x. PMID 9311400